CLINICAL TRIAL: NCT04568031
Title: A Phase I/II Randomized, Double-blind, Placebo-controlled Multicentre Study in Participants Aged 18 Years or Older to Determine the Safety and Immunogenicity of AZD1222, a Non-replicating ChAdOx1 Vector Vaccine, for the Prevention of COVID-19
Brief Title: Study of AZD1222 for the Prevention of COVID-19 in Japan
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D8111C00002
Record Dates: First submitted 2020-08-21; First posted 2020-09-29 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I (Active Comparator): Cohort C will include healthy participants aged 18 to 55 years. Cohort D will include healthy elderly participants aged ≥ 56 years. In Cohort D, the elderly population is further divided into 2 different age subgroups; aged 56 to 69 years (Subcohort D1) and aged ≥ 70 years (Subcohort D2). At least 30% of participants in Cohort D will be secured for participants with age ≥ 70 years.
  Interventions: Drug: AZD1222
- Part II (Placebo Comparator): Cohort C will include healthy participants aged 18 to 55 years. Cohort D will include healthy elderly participants aged ≥ 56 years. In Cohort D, the elderly population is further divided into 2 different age subgroups; aged 56 to 69 years (Subcohort D1) and aged ≥ 70 years (Subcohort D2). At least 30% of participants in Cohort D will be secured for participants with age ≥ 70 years.
  Interventions: Drug: 0.9% (w/v) saline

INTERVENTIONS:
Drug: AZD1222 — For subjects in part 1 will have that route of Administration as Intramuscular, 5 × 1010 vp (nominal, ± 1.5 × 1010 vp) on V2
  Arms: Part I
Drug: 0.9% (w/v) saline — For subjects in placebo will have that route of Administration as Intramuscular 0.9% (w/v) saline on V2 and V6.
  Arms: Part II

SUMMARY:
The COVID-19 pandemic has caused major disruption to healthcare systems with significant socioeconomic impacts. Currently, there are no licensed preventions available against COVID-19 and accelerated vaccine development is urgently needed. A safe and effective vaccine for COVID 19 prevention would have significant global public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 55 years (Cohort A and C), aged 56 to 69 years (Subcohorts B1 and D1), or aged ≥ 70 years (Subcohorts B2 and D2)

Exclusion Criteria:

1. Known past laboratory-confirmed SARS-CoV-2 infection
2. Positive SARS-CoV-2 RT PCR test at screening
3. Seropositivity to SARS-CoV-2 at screening.
4. Significant infection or other illness, including fever > 37.8°C on the day prior to or day randomization
5. History of Guillain-Barré syndrome
6. Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting ≤ 14 days)
7. History of allergy to any component of the vaccine
8. Any history of angioedema
9. Any history of anaphylaxis
10. Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and uterine cervical carcinoma in situ)
11. History of serious psychiatric condition likely to affect participation in the study
12. Bleeding disorder (eg, factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
13. Suspected or known current alcohol or drug dependency
14. Any other significant disease, disorder or finding which may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study or impair interpretation of the study data
15. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-08-23 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Research Site, Fukuoka
  - Research Site, Hachioji-shi
  - Research Site, Minatoku
  - Research Site, Sumida-ku
  - Research Site, Toshima-ku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ishikawa K, Nascimento MC, Asano M, Hirata H, Itoh Y, Kelly EJ, Matsui A, Olsson U, Shoemaker K, Green J. One year safety and immunogenicity of AZD1222 (ChAdOx1 nCoV-19): Final analysis of a randomized, placebo-controlled phase 1/2 trial in Japan. Vaccine. 2023 Jun 29;41(29):4199-4205. doi: 10.1016/j.vaccine.2023.05.015. Epub 2023 Jun 2. PMID 37271703
- [Derived] Asano M, Okada H, Itoh Y, Hirata H, Ishikawa K, Yoshida E, Matsui A, Kelly EJ, Shoemaker K, Olsson U, Vekemans J. Immunogenicity and safety of AZD1222 (ChAdOx1 nCoV-19) against SARS-CoV-2 in Japan: a double-blind, randomized controlled phase 1/2 trial. Int J Infect Dis. 2022 Jan;114:165-174. doi: 10.1016/j.ijid.2021.10.030. Epub 2021 Oct 22. PMID 34688944
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111C00002&attachmentIdentifier=1a2ff66f-3b83-44a1-a462-ce6df8a172c0&fileName=D933AC00001_-___Statistical_Analysis_Plan-redact.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111C00002&attachmentIdentifier=dca086b6-afe2-406b-9cc8-72a7105fc54a&fileName=d933ac00001-oncology-late-phase-master-csp-v8-redact.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111C00002&attachmentIdentifier=34124f37-74e8-428b-8905-fa99deb0154a&fileName=d933ac00001-study-synopsis-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I/II study was conducted in healthy, severe acute respiratory syndrome-coronavirus 2 (SARS-CoV-2) naïve participants at 5 study centers in Japan. First participant was randomized on 23 August 2020 and final data cut-off (DCO) date was 17 January 2022.
Pre-assignment Details: The study had a screening period (14 days), followed by vaccination and follow-up period (up to 365 days). The study consists of 2 cohorts (Cohort C and Cohort D) with different age populations. The Cohort C included participants aged 18 to 55 years and Cohort D included participants aged >= 56 years. A total of 256 participants were randomized in a 3:1 ratio to receive AZD1222 or placebo.
Groups:
- Cohort C: AZD1222: Participants were randomized to receive 2 intramuscular (IM) doses of either 5*10^10 viral particles (vp) (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Cohort C: Placebo; Cohort D: Placebo: Participants were randomized to receive 2 IM doses of placebo matching with AZD1222 on Days 1 and 29.
- Cohort D: AZD1222: Participants were randomized to receive 2 IM doses of either 5*10^10 vp (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
Period: Overall Study
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Started | 96 | 32 | 96 | 32
Participants Received 1 Vaccination | 96 | 32 | 96 | 32
Participants Received 2 Vaccinations | 84 | 30 | 92 | 31
Completed | 93 | 32 | 91 | 31
Not Completed | 3 | 0 | 5 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The Total vaccinated analysis set (TVS) included all participants who received at least 1 dose of study vaccination.
Groups:
- Cohort C: AZD1222; Cohort D: AZD1222: Participants were randomized to receive 2 IM doses of either 5*10^10 vp (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Total: Total of all reporting groups
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo | Total
Number analyzed (Participants) | 96 | 32 | 96 | 32 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 96 | 32 | 51 | 14 | 193
  >=65 years | 0 | 0 | 45 | 18 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 8 | 40 | 14 | 87
  Male | 71 | 24 | 56 | 18 | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 96 | 32 | 96 | 32 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 96 | 32 | 96 | 32 | 256

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroresponse to the Spike (S) Antigen of AZD1222 as Measured by Meso Scale Discovery (MSD) Serology Assay
Description: Seroresponse is a binary outcome where a success is when the fold rise in titers compared with baseline is >= 4. The fold rise in titers was calculated as the ratio of the post-vaccination titer level to the baseline titer level. The percentage of participants with a post-vaccination seroresponse (>= 4-fold rise in titers from Day 1 baseline value to Day 57) to the S antigen of AZD1222 as measured by MSD serology assay is reported.
Time Frame: Baseline (Day 1) and Day 57
Population: The Fully vaccinated analysis set (FVS) for immunogenicity included all participants in the TVS who received 2 study vaccinations and had no important protocol deviations judged to have the potential to interfere with the generation or interpretation of immune responses. Only participants evaluated for seroresponse at Day 57 are reported. Participants with seroresponse to nucleocapsid antibodies by MSD serology assay at post-baseline up to Day 57 were excluded from this analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 83 | 29 | 91 | 31
percentage of participants | 100.0 | 0.0 | 100.0 | 0.0
Statistical Analysis 1: Comparison: Cohort C: AZD1222 vs Cohort C: Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort D: AZD1222 vs Cohort D: Placebo; Test type: Superiority; p < 0.001, Fisher Exact

2. Primary Outcome: Number of Participants With Local Solicited Adverse Events (AE)
Description: Solicited AEs are local or systemic predefined AEs for reactogenicity assessment. Participants were given an axillary thermometer, tape measure, and access to app for the solicited AE eDiary, with instructions on use, along with the emergency 24-hour telephone number to contact the on-call study physician if needed. Participants were instructed to record for 7 days following administration of each dose of AZD1222, the timing and severity of local and systemic solicited AEs, if applicable, and whether medication was taken to relieve the symptoms.
Time Frame: From Day 1 up to 7 days post each dose of study vaccination, approximately 14 days
Population: The TVS included all participants who received at least 1 dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 96 | 32 | 96 | 32
Participants
  After first vaccination | 70 | 4 | 46 | 2
  After second vaccination: number analyzed (Participants) | 84 | 30 | 92 | 31
  After second vaccination | 37 | 3 | 36 | 0
  After any vaccination | 74 | 5 | 53 | 2

3. Primary Outcome: Number of Participants With Systemic Solicited AEs
Description: as for outcome 2
Time Frame: From Day 1 up to 7 days post each dose of study vaccination, approximately 14 days
Population: The TVS included all participants who received at least 1 dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 96 | 32 | 96 | 32
Participants
  After first vaccination | 65 | 6 | 41 | 3
  After second vaccination: number analyzed (Participants) | 84 | 30 | 92 | 31
  After second vaccination | 30 | 7 | 24 | 3
  After any vaccination | 68 | 11 | 47 | 5

4. Primary Outcome: Number of Participants With AEs, Serious AEs (SAE) and Adverse Event of Special Interest (AESI) Occurring Post Each Dose of Study Vaccination
Description: An AE is the development of any untoward medical occurrence in a clinical study participant administered medicinal product and which does not necessarily have a causal relationship with this medicinal product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is an AE occurring during any study phase that fulfils one or more of the following criteria: death; immediately life-threatening; in-participant hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital abnormality or birth defect; an important medical event. The AESIs were events of scientific and medical interest specific to the further understanding of the study vaccination safety profile and required close monitoring and rapid communication by the investigators to the sponsor.
Time Frame: From Day 1 up to 28 days post each dose of study vaccination, approximately 57 days
Population: The TVS included all participants who received at least 1 dose of study vaccination. Unsolicited AEs that started after the inoculation of non-study coronavirus disease 2019 vaccine were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 96 | 32 | 96 | 32
Participants
  AEs | 28 | 4 | 22 | 9
  SAEs | 0 | 1 | 3 | 1
  AESIs | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters
Description: Clinical laboratory values were evaluated for each laboratory parameter as applicable including hematology and clinical chemistry. The baseline was defined as the last non-missing measurement taken prior to the first dose of study vaccination (including unscheduled measurements, if any).
Time Frame: From Day 1 up to 28 days post each dose of study vaccination, approximately 57 days
Population: The TVS included all participants who received at least 1 dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 96 | 32 | 96 | 32
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Seroresponse to the Receptor-Binding Domain (RBD) Antigen of AZD1222 as Measured by MSD Serology Assay
Description: Seroresponse is a binary outcome where a success is when the fold rise in titers compared with baseline is >= 4. The fold rise in titers was calculated as the ratio of the post-vaccination titer level to the baseline titer level. The percentage of participants with a post-vaccination seroresponse (>= 4-fold rise in titers from Day 1 baseline value to Day 57) to the RBD antigen of AZD1222 as measured by MSD serology assay is reported.
Time Frame: Baseline (Day 1) and Day 57
Population: The FVS for immunogenicity included all participants in the TVS who received 2 study vaccinations and had no important protocol deviations judged to have the potential to interfere with the generation or interpretation of immune responses. Only participants evaluated for seroresponse at Day 57 are reported. Participants with seroresponse to nucleocapsid antibodies by MSD serology assay at post-baseline up to Day 57 were excluded from this analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 83 | 29 | 91 | 31
percentage of participants | 100.0 | 0.0 | 100.0 | 0.0
Statistical Analysis 1: Comparison: Cohort C: AZD1222 vs Cohort C: Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort D: AZD1222 vs Cohort D: Placebo; Test type: Superiority; p < 0.001, Fisher Exact

7. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 S and RBD Antibodies as Measured by MSD Serology Assay
Description: The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titer/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titer, where 'n' is the number of participants with titer information.
Time Frame: Baseline (Day 1) and Days 15, 29, 43, 57, 183, and 365
Population: The FVS for immunogenicity included all participants in the TVS who received 2 study vaccinations and had no important protocol deviations judged to have the potential to interfere with the generation or interpretation of immune responses. Participants with seroresponse to nucleocapsid antibodies by MSD serology assay at post-baseline up to Day 57 were excluded from this analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: arbitrary units per milliliter (AU/mL)
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 83 | 29 | 91 | 31
arbitrary units per milliliter (AU/mL)
  S Antibody Titer: Baseline (Day 1) | 62.18 [48.136 to 80.310] | 46.00 [32.713 to 64.672] | 39.06 [31.824 to 47.931] | 39.87 [24.214 to 65.662]
  S Antibody Titer: Day 15 | 2520.37 [1868.317 to 3399.988] | 43.70 [31.600 to 60.426] | 999.28 [751.737 to 1328.342] | 39.24 [24.016 to 64.105]
  S Antibody Titer: Day 29 | 7971.03 [6278.011 to 10120.625] | 42.66 [30.843 to 58.993] | 6720.46 [5361.399 to 8424.022] | 40.03 [24.956 to 64.223]
  S Antibody Titer: Day 43 | 17708.74 [14671.831 to 21374.262] | 41.61 [29.411 to 58.879] | 15594.37 [12792.879 to 19009.367] | 37.89 [23.025 to 62.344]
  S Antibody Titer: Day 57 | 14986.27 [12455.149 to 18031.758] | 44.24 [31.816 to 61.507] | 12824.27 [10516.280 to 15638.797] | 38.75 [23.604 to 63.618]
  S Antibody Titer: Day 183: number analyzed (Participants) | 82 | 26 | 90 | 31
  S Antibody Titer: Day 183 | 4454.01 [3503.969 to 5661.645] | 53.28 [36.416 to 77.945] | 3424.65 [2758.191 to 4252.152] | 45.89 [28.326 to 74.347]
  S Antibody Titer: Day 365: number analyzed (Participants) | 80 | 3 | 86 | 4
  S Antibody Titer: Day 365 | 3691.12 [2468.353 to 5519.626] | 760.64 [0.002 to 266254529.058] | 2691.98 [1910.675 to 3792.785] | 116.38 [0.611 to 22179.458]
  RBD Antibody Titer: Baseline (Day 1) | 122.62 [106.105 to 141.715] | 114.89 [96.952 to 136.148] | 105.41 [100.326 to 110.752] | 119.83 [97.625 to 147.077]
  RBD Antibody Titer: Day 15 | 945.33 [678.340 to 1317.392] | 116.04 [96.504 to 139.521] | 430.65 [329.174 to 563.418] | 118.91 [97.844 to 144.520]
  RBD Antibody Titer: Day 29 | 6466.23 [5026.530 to 8318.284] | 115.39 [96.817 to 137.518] | 5616.00 [4468.764 to 7057.759] | 116.63 [94.796 to 143.491]
  RBD Antibody Titer: Day 43 | 20719.36 [17079.781 to 25134.511] | 114.43 [97.164 to 134.766] | 17677.04 [14383.279 to 21725.058] | 123.20 [100.706 to 150.715]
  RBD Antibody Titer: Day 57 | 16775.12 [13921.806 to 20213.221] | 114.54 [97.063 to 135.156] | 14094.42 [11437.864 to 17367.992] | 116.24 [96.030 to 140.713]
  RBD Antibody Titer: Day 183: number analyzed (Participants) | 82 | 26 | 90 | 31
  RBD Antibody Titer: Day 183 | 4245.22 [3309.128 to 5446.106] | 111.24 [98.273 to 125.916] | 3354.78 [2646.741 to 4252.239] | 127.71 [95.347 to 171.052]
  RBD Antibody Titer: Day 365: number analyzed (Participants) | 80 | 3 | 86 | 4
  RBD Antibody Titer: Day 365 | 3550.69 [2296.498 to 5489.828] | 1520.17 [0.014 to 169886733.576] | 2643.76 [1811.827 to 3857.686] | 304.93 [9.346 to 9948.763]

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 S and RBD Antibodies as Measured by MSD Serology Assay
Description: The fold rise was calculated as the ratio of the post-vaccination titer level to the baseline titer level, where baseline was defined as the last measurement taken before the first dose of study vaccination. The GMFR was calculated as anti-logarithm of Σ (log base 2 transformed (post-vaccination titer/ pre-vaccination titer)/n). Where 'n' is the number of participants with titer information.
Time Frame: Baseline (Day 1) and Days 15, 29, 43, 57, 183, and 365
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 83 | 29 | 91 | 31
ratio
  S Antibody Titer: Day 15 | 40.54 [30.451 to 53.962] | 0.95 [0.863 to 1.046] | 25.59 [18.465 to 35.453] | 0.98 [0.865 to 1.119]
  S Antibody Titer: Day 29 | 128.20 [97.728 to 168.179] | 0.93 [0.841 to 1.023] | 172.07 [128.206 to 230.951] | 1.00 [0.869 to 1.161]
  S Antibody Titer: Day 43 | 284.82 [217.685 to 372.656] | 0.90 [0.814 to 1.006] | 399.28 [295.200 to 540.068] | 0.95 [0.842 to 1.072]
  S Antibody Titer: Day 57 | 241.03 [183.977 to 315.781] | 0.96 [0.881 to 1.050] | 328.36 [243.794 to 442.254] | 0.97 [0.858 to 1.100]
  S Antibody Titer: Day 183: number analyzed (Participants) | 82 | 26 | 90 | 31
  S Antibody Titer: Day 183 | 70.49 [51.130 to 97.171] | 1.11 [0.920 to 1.344] | 88.17 [65.621 to 118.464] | 1.15 [1.021 to 1.298]
  S Antibody Titer: Day 365: number analyzed (Participants) | 80 | 3 | 86 | 4
  S Antibody Titer: Day 365 | 59.15 [37.619 to 93.012] | 25.12 [0.000 to 26524735.936] | 70.56 [47.647 to 104.486] | 4.18 [0.042 to 416.314]
  RBD Antibody Titer: Day 15 | 7.71 [5.690 to 10.445] | 1.01 [0.995 to 1.025] | 4.09 [3.140 to 5.315] | 0.99 [0.972 to 1.013]
  RBD Antibody Titer: Day 29 | 52.73 [40.850 to 68.070] | 1.00 [0.985 to 1.024] | 53.28 [42.740 to 66.413] | 0.97 [0.915 to 1.035]
  RBD Antibody Titer: Day 43 | 168.97 [134.602 to 212.105] | 1.00 [0.983 to 1.009] | 167.70 [137.013 to 205.253] | 1.03 [0.966 to 1.095]
  RBD Antibody Titer: Day 57 | 136.80 [109.050 to 171.614] | 1.00 [0.992 to 1.002] | 133.71 [108.961 to 164.080] | 0.97 [0.911 to 1.033]
  RBD Antibody Titer: Day 183: number analyzed (Participants) | 82 | 26 | 90 | 31
  RBD Antibody Titer: Day 183 | 34.54 [26.040 to 45.820] | 0.96 [0.891 to 1.023] | 31.81 [25.259 to 40.071] | 1.07 [0.888 to 1.279]
  RBD Antibody Titer: Day 365: number analyzed (Participants) | 80 | 3 | 86 | 4
  RBD Antibody Titer: Day 365 | 28.76 [18.123 to 45.629] | 14.90 [0.000 to 1665556.212] | 25.03 [17.383 to 36.049] | 2.99 [0.092 to 97.537]

9. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Neutralizing Antibodies (nAb) of AZD1222 as Measured by Pseudo-Neutralization Assay
Description: Seroresponse is a binary outcome where a success is when the fold rise in titers compared with baseline is >= 4. The fold rise in titers was calculated as the ratio of the post-vaccination titer level to the baseline titer level. The percentage of participants with a post-vaccination seroresponse (>= 4-fold rise in titers from Day 1 baseline value to Day 57) to SARS-CoV-2 nAb of AZD1222 as measured by pseudo-neutralization assay is reported.
Time Frame: Baseline (Day 1) and Day 57
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 80 | 29 | 86 | 30
percentage of participants | 67.5 | 0.0 | 57.0 | 0.0
Statistical Analysis 1: Comparison: Cohort C: AZD1222 vs Cohort C: Placebo; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort D: AZD1222 vs Cohort D: Placebo; Test type: Superiority; p < 0.001, Fisher Exact

10. Secondary Outcome: GMTs for SARS-CoV-2 nAb as Measured by Pseudo-Neutralization Assay
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Days 29, 57, 183, and 365
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 83 | 29 | 91 | 31
AU/mL
  Baseline (Day 1) | 20.84 [19.206 to 22.604] | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the lower limit of quantification (LLOQ) was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and upper limit of quantification (ULOQ) is 787339 AU/mL. | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 20.82 [19.175 to 22.616]
  Day 29: number analyzed (Participants) | 75 | 29 | 85 | 31
  Day 29 | 67.26 [50.689 to 89.249] | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 46.11 [36.577 to 58.132] | 21.07 [18.947 to 23.422]
  Day 57: number analyzed (Participants) | 80 | 29 | 86 | 30
  Day 57 | 107.30 [84.198 to 136.741] | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 90.00 [70.051 to 115.618] | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL.
  Day 183: number analyzed (Participants) | 81 | 26 | 88 | 31
  Day 183 | 31.14 [24.679 to 39.281] | 20.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 28.91 [24.717 to 33.810] | 20.54 [19.448 to 21.703]
  Day 365: number analyzed (Participants) | 76 | 3 | 83 | 4
  Day 365 | 43.16 [28.917 to 64.428] | 97.03 [0.109 to 86708.084] | 32.44 [24.376 to 43.159] | 25.40 [11.875 to 54.316]

11. Secondary Outcome: GMFR for SARS-CoV-2 nAb as Measured by Pseudo-Neutralization Assay
Description: as for outcome 8
Time Frame: Baseline (Day 1) and Days 29, 57, 183, and 365
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 81 | 29 | 88 | 31
ratio
  Day 29: number analyzed (Participants) | 75 | 29 | 85 | 31
  Day 29 | 3.21 [2.469 to 4.184] | 1.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 2.31 [1.829 to 2.907] | 1.01 [0.988 to 1.036]
  Day 57: number analyzed (Participants) | 80 | 29 | 86 | 30
  Day 57 | 5.14 [4.066 to 6.503] | 1.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 4.50 [3.503 to 5.781] | 1.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL.
  Day 183: number analyzed (Participants) | 81 | 26 | 88 | 31
  Day 183 | 1.49 [1.186 to 1.879] | 1.00 [NA to NA] — Lower and upper limit of confidence interval was not evaluable due to below the level of detection. A titer value measured below the LLOQ was imputed to a value that is half of the LLOQ in summaries and analyses. The value of LLOQ is 40 AU/mL and ULOQ is 787339 AU/mL. | 1.45 [1.236 to 1.690] | 0.99 [0.960 to 1.014]
  Day 365: number analyzed (Participants) | 76 | 3 | 83 | 4
  Day 365 | 2.06 [1.379 to 3.088] | 4.85 [0.005 to 4335.404] | 1.62 [1.219 to 2.158] | 1.27 [0.594 to 2.716]

12. Secondary Outcome: Number of Participants With SAEs and AESIs Occurring Throughout the Study
Description: An SAE is an AE occurring during any study phase that fulfils one or more of the following criteria: death; immediately life-threatening; in-participant hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital abnormality or birth defect; an important medical event. The AESIs were events of scientific and medical interest specific to the further understanding of the study vaccination safety profile and required close monitoring and rapid communication by the investigators to the sponsor.
Time Frame: From Day 1 up to final DCO of 17 January 2022, up to a maximum of 365 days
Population: The TVS included all participants who received at least 1 dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: AZD1222 | Cohort C: Placebo | Cohort D: AZD1222 | Cohort D: Placebo
Number analyzed (Participants) | 96 | 32 | 96 | 32
Participants
  SAEs | 0 | 2 | 3 | 1
  AESIs | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs are reported from first administration of study vaccination up to final DCO of 17 January 2022, up to a maximum of 365 days
Description: The TVS included all participants who received at least 1 dose of study vaccination.
Groups:
- Cohorts C + D: AZD1222: Participants were randomized to receive 2 IM doses of either 5*10^10 vp (nominal, ± 1.5*10^10 vp) AZD1222 on Days 1 and 29.
- Cohorts C + D: Placebo: Participants were randomized to receive 2 IM doses of placebo matching with AZD1222 on Days 1 and 29.
Arm/Group | Cohorts C + D: AZD1222 | Cohorts C + D: Placebo
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/64
Serious Adverse Events (participants affected / at risk) | 3/192 | 3/64
Other Adverse Events (participants affected / at risk) | 11/192 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts C + D: AZD1222 (N=192) | Cohorts C + D: Placebo (N=64)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts C + D: AZD1222 (N=192) | Cohorts C + D: Placebo (N=64)
Tenderness (General disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04568031/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT04568031/SAP_001.pdf